CLINICAL TRIAL: NCT02826447
Title: ANRS 12320 IMMHoTHep : Investigative Mathematical Modeling of Hospital Transmission of Hepatitis C
Brief Title: Investigative Mathematical Modeling of Hospital Transmission of Hepatitis C
Acronym: IMMHoTHep
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Conservatoire national des Arts et Métiers (Other); Ain Shams University (Other); Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: ANRS 12320
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Exposure to Hepatitis C Virus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples With DNA — Blood sample (5mL)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: 500 patients who are going to be hospitalized for at least 24 hours at Ain Shams University Teaching Hospital in the following departments: surgery, internal medicine, gynecology/obstetrics and toxicology.
- Healthcare workers: 50 healthcare workers working at Ain Shams University Teaching Hospital in the following departments: surgery, internal medicine, gynecology/obstetrics and toxicology.

SUMMARY:
This project is a prospective observational cohort study to quantify the risk of acquiring Hepatitis C virus (HCV) infection for patients and healthcare workers in Ain Shams University Teaching Hospital, Cairo, Egypt through: 1) identifying typical patient trajectories within the hospital; and 2) assessing the ward-specific risk based on the type and number of procedures performed and the prevalence of HCV viremia in patients within each ward.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) is a blood-borne virus and its major route of transmission include blood transfusion, medical injection and procedure, and injecting drug use. In Egypt, the origin of the HCV epidemic has been attributed to a mass treatment of schistosomiasis between 1960 and 1984, when intravenous injections with antimony salts were given to 3-5 million people older than 6 years of age. Insufficient sterilization of needles and syringes was considered to be responsible for HCV transmission at that time. In order to control the spread of HCV in Egypt, the Egyptian Ministry of Health and Population established the National Committee for the Control of Viral Hepatitis. By 2008, this committee developed a National Control Strategy for Viral Hepatitis which has recommended prevention and education campaigns targeting general population and also healthcare workers (HCW). In their occupational environment, HCWs are frequently exposed to multiple blood-borne pathogens, including HCV. Several risk factors for HCV acquisition among patients and HCWs within a hospital ward have been identified, including a high prevalence of HCV infection in the ward, understaffing, workplace characteristic, and human factors such as inexperience or unfamiliar with equipment. However, to the investigators' knowledge, the overall risk of HCV acquisition associated with hospital stay has never been evaluated in Egypt. Also, control measures to reduce the risk of HCV transmission in hospital settings, based on a global assessment of healthcare provider logistics and performance, have never been proposed in Egypt.

In this project, the investigators assume that HCV will be transmitted to both hospital staff and patients. Given the slow dynamics of the HCV epidemic, the investigators further hypothesize that, in the short term, the prevalence of HCV viremia among patients will be constant. Therefore, the investigators are led to conclude that HCV transmission risk may be inferred from a detailed description of individual trajectories of patients or staff within the hospital.

ELIGIBILITY:
Inclusion Criteria for patients:

* Aged 21 years or older
* Staying in the hospital more than 24 hours
* Provided a written informed consent to participate

Inclusion Criteria for healthcare workers:

* Aged 21 or older
* Provided a written informed consent to participate

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 500 patients staying at least 24 hours in one of the following departments of the Ain Shams University Teaching Hospital: surgery, internal medicine, gynecology/obstetrics and toxicology.
  50 healthcare workers working in one of departments cited above.
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Per-day risk of HCV acquisition for a hospitalized patient | 1 day
  Per-day risk of HCV acquisition for a hospitalized patient
Per-week risk of HCV acquisition for a healthcare worker through occupational blood exposure | 1 week
  Per-week risk of HCV acquisition for a healthcare worker through occupational blood exposure

SECONDARY OUTCOMES:
Estimation of the number of HCV acquisitions among patients and HCWs prevented over a 1-year period following the implementation of various control strategies, using a mathematical modeling approach | 1 year
  Estimation of the number of HCV acquisitions among patients and HCWs prevented over a 1-year period following the implementation of various control strategies,

CONTACTS AND LOCATIONS:
Overall Officials: Laura Temime, Professor, Principal Investigator — Conservatoire national des Arts et Métiers; Wagida Anwar, Professor, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Teaching Hospital, Cairo, Egypt